CLINICAL TRIAL: NCT01871649
Title: A Randomized, Double-blind, Placebo-controlled Trial of Golimumab+Methotrexate Versus Methotrexate Alone in Methotrexate-naïve Patients With Psoriatic Arthritis
Brief Title: Initial Treatment With Golimumab in Early PsA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, D.L.P. Baeten, prof. dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AMC_ 42670_PsA_Golimumab
Record Dates: First submitted 2013-01-07; First posted 2013-06-07 (Estimated); Last update posted 2018-11-26 (Actual); Status verified 2018-11

CONDITIONS: Psoriatic Arthritis
Keywords: psoriatic arthritis; golimumab; methotrexate; minimal disease activity; safety; withdrawal
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — golimumab; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- methotrexate (Active Comparator): methotrexate is the active comparator, it will be compared to golimumab + methotrexate
  Interventions: Drug: methotrexate
- golimumab and methotrexate (Experimental): The combination of golimumab en methotrexate will be compared to methotrexate alone.
  Interventions: Drug: golimumab

INTERVENTIONS:
Drug: golimumab — golimumab 50mg subcutaneous injections (in combination with methotrexate), once a month, for a period of 22 weeks
  Other Names: simponi
  Arms: golimumab and methotrexate
Drug: methotrexate — Methotrexate will be started at a dosage of 15 mg/week orally and, if well tolerated, increased to 20mg/week at week 4 and 25mg/week at week 8 of the trial. If well tolerated, the maximum dose of 25 mg/week will be sustained until end of study (week 50). Folic acid 5 mg/week will be administered orally one day after the MTX intake.
  Arms: methotrexate

SUMMARY:
The investigators will perform a 22-week randomized, double-blind, placebo-controlled trial of golimumab + methotrexate (MTX) versus methotrexate alone in methotrexate-naïve patients with Psoriatic Arthritis (PsA). Afterwards, a 28 week open label phase with methotrexate alone is started. Golimumab will be discontinued.

Hypotheses:

First, the investigators hypothesize that initiation of a combination therapy with golimumab + MTX will be safe and superior to MTX alone in MTX-naïve PsA patients, as assessed by the percentage of patients achieving Disease Activity Score (the investigators hypothesize that more patients with the early combination treatment will respond (according to Disease Activity Score (DAS), American college of Rheumatology (ACR), or Psoriatic Arthritis Response Criteria (PsARC) responses) and achieve a state of Low Disease Activity (LDA) or Minimal Disease Activity (MDA) than patients on MTX alone.

Third, the investigators hypothesize that a significant proportion of the patients will continue to benefit from this early aggressive treatment initiation even after stopping golimumab treatment.

ELIGIBILITY:
Inclusion Criteria:

* Prior to any study procedure, voluntary written informed consent must be obtained, after the nature and purpose of this study were explained
* Patients should be between 18 and 70 years of age at time of consent
* Patients must have a diagnosis of PsA according to the Classification for psoriatic Arthritis (CASPAR) classification criteria (see Appendix 1).
* The patient must have an active disease as defined by 3 swollen and 3 tender joints.
* The use of a stable dose of concomitant nonsteroidal antiinflammatory drug (NSAIDs) and/or corticosteroids is allowed. The dose of corticosteroids should not exceed a prednisone equivalent of 10 mg/day and must be stable for at least 4 weeks prior to baseline. The dose of concomitant NSAIDs and corticosteroids should be kept stable during the whole study period.
* Patients are considered to be in generally good health based upon the result of a medical history, physical examination, laboratory profile, chest X-ray and electrocardiography (ECG).

Exclusion Criteria:

* Patient has a concomitant rheumatic condition other than PsA
* Positivity for rheumatoid factor (RF) or anti-cyclic citrullinated peptide (anti CCP) antibodies (ACPA)
* Current or previous use of methotrexate
* Current use of other Disease Modifying Antirheumatic drug (DMARDs) (sulphasalazine or leflunomide).
* Prior use of other DMARDs (sulphasalazine or leflunomide) within 3 months before baseline.
* Current or previous use of biologicals, including Tumor Necrosis Factor (TNF) blocking therapy
* Patient has active tuberculosis. A purified protein derivative (PPD) skin test and chest X-ray at screening should be negative (in case of latent tuberculosis, a patient may enter the study if prophylaxis with isoniazide is begun prior to administration of study medication). If a patient has an adequately treated tuberculosis in the past, he/she may enter the trial.
* Patient has received an intra-articular injection with corticosteroids within 4 weeks prior to baseline.
* Patient has a malignancy (other than basal cell carcinoma of the skin) in the past 5 years
* Patients has a recent history of (or persistent) infection requiring hospitalization or antibiotic treatment within 4 weeks of baseline Patient has a significant history of cardiac, pulmonary, renal (glomerular filtration rate <40ml/min), hepatic (liver cirrhosis), hematological, neurological, metabolic or any other disease that may affect his/her participation in this study. This should be decided by the opinion of the investigator.
* All females of childbearing potential must use appropriate contraception, be postmenopausal or surgically sterile. A urine pregnancy-test beta-human chorion gonadotropin (Beta-HCG) will be performed at screening and has to be negative.
* Subject is pregnant or a breastfeeding woman
* Liver disease or liver injury as indicated by abnormal liver function tests such as Alanine aminotransferase (ALT), Aspartate aminotransferase (AST), gammaglutamyl transpeptidase (GGT), alkaline phosphatase, or serum bilirubin. The Investigator should be guided by the following criteria: Any single parameter may not exceed 2 x upper limit of normal (ULN).

A single parameter elevated up to and including 2 x ULN should be rechecked once more if elevation levels are found clinically relevant according to the physician, at least prior to enrolment.

- Patient is, in the opinion of the investigator, unable to comply with the requirements of the study protocol or is unsuitable for the study for any reason.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Percentage of patients achieving DAS remission response criteria | week 22
  1. To demonstrate that golimumab + MTX is superior to MTX alone in achieving DAS remission in MTX naïve PsA patients at week 22
  DAS = Disease activity score, remission is defined as a DAS < 1.6
Number of Participants with Adverse Events | week 22
  Number of patients with(severe) adverse events (and type) during the study period.
  Safety will be monitored during the study period by laboratory tests and physical examination.

SECONDARY OUTCOMES:
Number of patients fulfilling Minimal Disease activity criteria and other outcome measurements | week 22
  To demonstrate that golimumab + MTX is superior to MTX alone as assessed by DAS, ACR and PsARC responses, as well as by achievement of low disease activity (LDA, as defined by DAS<2.4) and minimal disease activity (MDA, as defined by Coates et al, Ann Rheum Dis 2010). Also the Maastricht Ankylosing Spondylitis Enthesitis Score (MASES) score and Psoriasis Area Severity Index (PASI) score will be determined in MTX naïve PsA patients at week 22.

OTHER OUTCOMES:
Efficacy after withdrawing anti-TNF | week 50
  To demonstrate that initial treatment of MTX naïve patients with golimumab + MTX is superior to MTX alone to maintain DAS (disease activity score) remission, LDA (Low Disease Activity) and MDA over time (up to week 50) after withdrawing golimumab.

CONTACTS AND LOCATIONS:
Overall Officials: Dominique LP Baeten, Prof. dr. MD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (2):
- Netherlands (2):
  - Reade, Amsterdam, North Holland
  - Academic Medical Center/University of Amsterdam, Amsterdam, North Holland

REFERENCES:
- [Derived] de Jong HMY, van Mens LJJ, Nurmohamed MT, Kok MR, van Kuijk AWR, Baeten DLP, van de Sande MGH. Sustained remission with methotrexate monotherapy after 22-week induction treatment with TNF-alpha inhibitor and methotrexate in early psoriatic arthritis: an open-label extension of a randomized placebo-controlled trial. Arthritis Res Ther. 2019 Sep 14;21(1):208. doi: 10.1186/s13075-019-1998-4. PMID 31521192
- [Derived] van Mens LJJ, de Jong HM, Fluri I, Nurmohamed MT, van de Sande MGH, Kok M, van Kuijk AWR, Baeten D. Achieving remission in psoriatic arthritis by early initiation of TNF inhibition: a double-blind, randomised, placebo-controlled trial of golimumab plus methotrexate versus placebo plus methotrexate. Ann Rheum Dis. 2019 May;78(5):610-616. doi: 10.1136/annrheumdis-2018-214746. Epub 2019 Feb 26. PMID 30808625